CLINICAL TRIAL: NCT03374228
Title: A Study to Evaluate the Absolute Bioavailability of BMS-986205 Tablet Formulation
Brief Title: A Study to Evaluate the Bioavailability of BMS-986205
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CA017-060; 2017-003100-51 (EudraCT Number)
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — linrodostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986205 (Experimental): Single oral dose of BMS-986205 tablet on the morning of Day 1 followed by a 15-minute infusion of [13C]BMS-986205 solution for intravenous administration starting 01:45 hours after the oral dose administration
  Interventions: Drug: BMS-986205

INTERVENTIONS:
Drug: BMS-986205 — Specified Dose on Specified Days

SUMMARY:
Assess the absolute bioavailability of a tablet formulation of BMS-986205 following simultaneous oral administration of BMS-986205 and intravenous infusion of [13C]BMS-986205 solution for intravenous administration in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18.0 to 32.0 kg/m2, inclusive
* Must have normal renal function demonstrated by an estimated glomerular filtration rate, calculated by Chronic Kidney Disease Epidemiology Collaboration formula
* Women must not be of childbearing potential (cannot become pregnant)

Exclusion Criteria:

* Women who are of childbearing potential or breastfeeding
* Any significant acute or chronic medical illness
* Active tuberculosis (TB) requiring treatment or documented latent TB at screening

Other protocol defined inclusion / exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
Absolute oral bioavailability (F) | Up to 15 days
  Measured by plasma concentration

SECONDARY OUTCOMES:
Occurrence of adverse events (AEs) | Up to 15 days
  Safety and tolerability as measured by incidence of AEs
Occurrence of serious adverse events (SAEs) | Up to 15 days
  Safety and tolerability as measured by incidence of SAEs
Occurrence of adverse events (AEs) leading to discontinuation | Up to 15 days
  Safety and tolerability as measured by incidence of AEs leading to discontinuation
Number of participants with vital sign measurement abnormalities | Up to 15 days
Number of participants with electrocardiogram abnormalities | Up to 15 days
Number of participants with physical examination abnormalities | Up to 15 days
Number of participants with clinical laboratory test abnormalities | Up to 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Quotient Clinical, Nottingham, Ruddington Fields, United Kingdom

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS clinical trial educational resource — https://www.bmsstudyconnect.com/s/US/English/USenHome